CLINICAL TRIAL: NCT03318991
Title: Clinical Outcomes of Laser Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Fu-Shun Hsu, Doctoral student, Graduate Institute of Clinical Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTCH17001
Record Dates: First submitted 2017-10-16; First posted 2017-10-24 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Prostatic Hypertrophy
Keywords: thulium laser; GreenLight laser; laser therapy; resection of the prostate; prostate hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GreenLight laser (Active Comparator): 180W Greenlight laser is used for vaporesection of the prostate.
  Interventions: Procedure: Laser prostatectomy
- Thulium laser (Active Comparator): 200W Thulium laser is used for enucleation of the prostate.
  Interventions: Procedure: Laser prostatectomy

INTERVENTIONS:
Procedure: Laser prostatectomy — Patients with symptomatic benign prostate obstruction (BPO) will be assigned under randomisation to treat with GreenLight laser or thulium laser.

SUMMARY:
Benign prostate obstruction (BPO) can be treated with a range of laser treatments using different laser systems and applications. Transurethral laser treatment is considered to be an alternative treatment to transurethral resection of the prostate (TURP). The latest guidelines of the European Association of Urology recommend 532-nm GreenLight laser vaporisation of the prostate and thulium laser enucleation as alternatives to TURP. For further investigation of the efficacy of GreenLight and thulium laser in treating BPH, the investigators organize a prospective randomised control study. The investigators will enrol 100 patients with BPO, treated with either GreenLight laser or thulium laser prostatectomy, and compare their safety and efficacy.

DETAILED DESCRIPTION:
80 patients with symptomatic benign prostate obstruction (BPO) will be assigned under randomization to treat with GreenLight laser or thulium laser. Randomization is performed by free randomization software.

Inclusion criteria are patient age greater than 50 years, maximum flow rate (Qmax) < 15 ml/second and an International Prostate Symptom Score (IPSS) ≥ 10. The data for the quality-of-life questionnaire (QoL) and transrectal ultrasound measurement of the prostate (TRUS) are obtained preoperatively.

Exclusion criteria are known prostate cancer, bladder cancer, previous transurethral surgery, interstitial cystitis and neurogenic bladder confirmed after urodynamic studies. The use of anticoagulants or platelet aggregation inhibition and urinary retention under catheterization is not a criterion for study exclusion. The local institutional review board committee has approved the study as well as the data analysis.

Sample size The sample size was determined based on an expected mean IPSS of 5.8 ± 2.6 at 1-year followup. The investigators considered a change of deference of IPSS ≤ 2 as an accepted equivalence between the two groups. The sample size was calculated to be at least 21 patients in each group with α=0.05, β=0.80 and a desired statistical power level of 80%. Considering the possibility of patients drop out or lost to followup, 40 patients will be enrolled in each arm. All measurement data will be presented as mean ± standard deviation.

Statistical analysis StataCorp Stata 15 was used for statistical analysis. The Fisher's exact test was applied to compare categorical variables; and the Student's t-test was used to compare quantitative variables between the two treatment groups. A mixed model with random effect and Bonferroni correction was applied to compare IPSS, QoL, Qmax, and PVR between two groups. A two-sided P-value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patient age greater than 50 years, maximum flow rate (Qmax) < 15 ml/second and an International Prostate Symptom Score (IPSS) ≥ 10.

Exclusion Criteria:

* Exclusion criteria are known prostate cancer, bladder cancer, previous transurethral surgery, interstitial cystitis and neurogenic bladder confirmed after urodynamic studies.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
IPSS at 1 year | 1 year
  The primary outcome measurement is International Prostate Symptom Score (IPSS) at 1 year. The minimum and maximum scores are 0 and 35. The higher score means worse symptoms.

SECONDARY OUTCOMES:
Maximal flow rate (Qmax) | 1 year
  Maximal uroflow rate at 1 year, compared with preoperative data
Quality-of-life questionnaire | 1 year
  QoL score at 1 year, compared with preoperative data; The score ranges from 0 (the best) to 6 (the worst).

CONTACTS AND LOCATIONS:
Locations (1):
- New Taipei City Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Result] Thomas JA, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Bachmann A. A Multicenter Randomized Noninferiority Trial Comparing GreenLight-XPS Laser Vaporization of the Prostate and Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Obstruction: Two-yr Outcomes of the GOLIATH Study. Eur Urol. 2016 Jan;69(1):94-102. doi: 10.1016/j.eururo.2015.07.054. Epub 2015 Aug 15. PMID 26283011
- [Result] Netsch C, Becker B, Tiburtius C, Moritz C, Becci AV, Herrmann TRW, Gross AJ. A prospective, randomized trial comparing thulium vapoenucleation with holmium laser enucleation of the prostate for the treatment of symptomatic benign prostatic obstruction: perioperative safety and efficacy. World J Urol. 2017 Dec;35(12):1913-1921. doi: 10.1007/s00345-017-2071-z. Epub 2017 Jul 11. PMID 28698991
- [Result] Zhao C, Yang H, Chen Z, Ye Z. Thulium Laser Resection Versus Plasmakinetic Resection of Prostates in the Treatment of Benign Prostate Hyperplasia: A Meta-Analysis. J Laparoendosc Adv Surg Tech A. 2016 Oct;26(10):789-798. doi: 10.1089/lap.2016.0044. Epub 2016 Aug 8. PMID 27500451